CLINICAL TRIAL: NCT03995485
Title: Evaluation of Efficacy and Safety of KW-136 Capsule Combined With Sofosbuvir Tablet for Treatment of Adult Chronic Hepatitis C: an Open-label, Multi-center, Phase 3 Study
Brief Title: KW-136 With Sofosbuvir for Chinese Adults With Chronic Hepatitis C
Acronym: KW-136_III
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kawin Technology Share-holding Co., Ltd. (Industry)
Collaborators: KawinGreen Biotech Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KYGL-2017-001; CTR20171654 (Registry Identifier: China Drug Trials)
Record Dates: First submitted 2019-06-20; First posted 2019-06-24 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Hepatitis C, Chronic
Keywords: Chronic hepatitis C; Hepatitis C virus; Eradication; KW-136; Sofosbuvir; Nonstructural protein 5A; Nonstructural protein 5B; Panogentypic regimen; Confirmatory study
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — Sofosbuvir

STUDY DESIGN:
Intervention Model Description: Single-arm, external (historic) control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KW-136+SOF (Experimental): Treatment-naive and experienced subjects were medicated with KW-136 capsules 60 mg once daily and fixed-dose (400 mg once daily) sofosbuvir tablets for 12 successive weeks.
  Interventions: Drug: KW-136 capsule; Drug: Sofosbuvir

INTERVENTIONS:
Drug: KW-136 capsule — KW-136 60 mg was provided in a single capsule of 60 mg.
  Other Names: Coblopasvir
Drug: Sofosbuvir — Sofosbuvir was provided in a single tablet of 400 mg.

SUMMARY:
This study aimed to confirm efficacy and safety of KW-136, an investigational anti-hepatitis C virus (HCV) drug, combined with sofosbuvir for treatment of naive and experienced adults chronically infected with HCV. Three hundred and sixty (360) non-cirrhotic and cirrhotic subjects were medicated with KW-136 60 mg daily and sofosbuvir 400 mg daily. The treatment course lasted 12 successive weeks; thereafter all the study participants entered into a 12-week treatment-free follow-up period and an additional 12-week extension treatment-free follow-up period.

DETAILED DESCRIPTION:
It is estimated that China has a population of over 10 million infected with HCV and also a highly variable HCV genotype geographic distribution. A simple, universal, non-genotype-specific treatment regimen is preferred for anti-HCV treatment in clinical practice and public health. KW-136 and sofosbuvir are potent anti-HCV agents targeting at different HCV proteins, namely, nonstructural protein 5A and 5B, respectively. The combination regimen of KW-136 and sofosbuvir is expected to completely suppress HCV replication in subjects chronically infected with HCV and achieve a sustained virologic response (SVR12), namely, HCV not detected or below a predefined limit in plasma, 12 or 24 weeks after cessation of treatment.

In a previous phase 2 exploratory study, an all-oral, ribavirin-free regiment of KW-136, an investigational HCV NS5A inhibitor, combined with sofosbuvir, demonstrated a ~99% SVR12 in treatment-naive adult subjects chronically infected with major genotypes of HCV found in China, including those with compensatory cirrhosis. This phase 3 study aimed to confirm the efficacy and safety of this combined regimen in a large scale of target patient population, including interferon-experienced subjects. This simple, uniform regimen is expected to be the solution to HCV eradication in China from the perspective of public health.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 70 years (both inclusive) at the time of informed consenting and of either sex
* with a body mass index (BMI) between 18 and 32 kg/m^2 (both inclusive)
* chronically infected with HCV, namely, with positive anti-HCV, HCV RNA or genotyping results at least six (6) months before the screening, or with a liver biopsy confirming chronic hepatitis at most twelve (12) months before the screening or within the screening period
* with anti-HCV positivity and at least once testing result with HCV RNA equaling to or above 10^4 IU/mL within the screening period
* with gentoype 1, 2, 3, 4, 5, 6, mixed, indeterminate or other genotype by the centralized laboratory genotyping
* no more than ten percent (10%) of the enrolled subjects having previously experienced interferon (defined as having received any regulatory agency approved or investigational interferon formulations, including pegylated and regular interferons at least six [6] months before the screening)
* having not previously experienced any other approved, investigational or unapproved direct antiviral agents against HCV of any source
* having not previously experienced oral or injective ribavirin within three (3) months before the screening
* no more than ten percent (10%) of the enrolled patients having advanced fibrosis or compensatory cirrhosis (as documented by liver transient elastography [FibroScan] within the screening period, or liver biopsy within twelve [12] months before the screening or within the screening period, with an evidence priority over FibroScan result and with the most recent biopsy prevailing in case of inconsistency between liver biopsy and FibroScan result), in accordance with the following definitions of liver disease: no advanced fibrosis or cirrhosis, with a liver stiffness modulus (LSM) below 9.6 kPa and/or F0-2 on fibrosis staging; advanced fibrosis, with a LSM equaling to or above 9.6 kPa but below 14.6 kPa and/or F3 on fibrosis staging; and cirrhosis, with a LSM equaling to or above 14.6 kPa and/or F4 on fibrosis staging
* women of childbearing potential (including postmenopausal women at or under 50 years of age) with negative blood pregnancy test results, and subjects of childbearing potential (including male subjects and their female partners) having no childbearing plan and consenting to voluntarily use effective contraceptive measures from the screening until six (6) months after the end of treatment
* lactating women consenting to discontinue nursing from the screening until six (6) months after the end of treatment
* voluntarily participating in this trial and being able to understand and sign the informed consent form

Exclusion Criteria:

* having previously experienced any investigational or experimental direct antiviral agents against HCV, including protease inhibitor, nonstructural protein (NS) 5A inhibitor or NS5B polymerase inhibitor, before the screening NS5B polymerase or NS5A inhibitors, before the screening
* having previously experienced interferon-based antiviral regimens within six (6) months before the screening
* having previously experienced oral or injective ribavirin within three (3) months before the screening
* having previously experienced any systemic potent immunomodulatory agents, such as steroids or thymosin alfa, excluding nasal, inhalational, topical steroids and/or others, for more than two (2) weeks within six (6) months before the screening, or expected to be exposed to these agents during the study period
* with hepatitis B virus surface antigen (HBsAg) or anti-human immunodeficient virus (HIV) positivity
* with evidence of decompensatory liver function, including but not limited to total serum bilirubin (TBIL) above twice (2) of the upper limit of normal (ULN), serum albumin (ALB) below 35 g/L or prothrombin activity (PTA) below 60% confirmed on repeated testing, previous or present history of ascites, upper gastrointestinal bleeding and/or hepatic encephalopathy, or with a liver function reserve of Child-Pugh class B or C
* with primary liver cancer confirmed or evidenced by serum alfa-fetoprotein (AFP) above 100 ng/ml or liver imaging study showing suspected nodules
* with a previous history of liver disease of other causes, including alcoholic liver disease, nonalcoholic steatohepatitis, drug-induced hepatitis, autoimmune hepatitis, Wilson disease or hemochromatosis
* with serum alanine aminotransferase (ALT) or asparate aminotransferase (AST) above ten (10) times of the ULN confirmed on repeated testing
* with white blood cell (WBC) count below 3×10^9 per liter, neutrophil count below 1.5×10^9 per liter (or below 1.25×10^9 per liter for cirrhotics), platelet count below 50×10^9 per liter, or hemoglobin below 100 g/L confirmed on repeated testing
* with serum creatinine clearance (CLcr) below 50 ml/min using the Cockcroft-Gault formula confirmed on repeated testing
* with poorly controlled diabetes mellitus (hemoglobin A1c [HbA1c] above 8.0% confirmed on repeated testing)
* with psychiatric or neurologic disorders, including previous or family history of psychiatric disorders (especially depression, depressive state, epilepsy or hysteria)
* with serious cardiovascular disorders, including uncontrolled hypertension (systolic blood pressure at or above 160 mmHg and/or diastolic blood pressure at or above 100 mmHg), heart insufficiency of New York Heart Association class III or above, history of myocardial infarction within six (6) months before the screening, history of percutaneous transluminal coronary angioplasty within six (6) months before the screening, unstable angina pectoris, or QTc interval (Fridericia correction formula QTc = QT×RR^-1/3) at or above 450 msec for males or 470 msec for females, second- or third-grade atrioventricular block or any other uncontrolled arrhythmias confirmed on repeated electrocardiography on screening
* with serious hematologic disorders, such as anemia, hemophilia and others
* with serious kidney diseases, such as chronic kidney disease, kidney insufficiency and others
* with serious gastrointestinal disorders, such as peptic ulcer, colitis and others
* with serious respirator disorders, such as active pulmonary tuberculosis, lung infection, chronic obstructive pulmonary disease, pulmonary interstitial disease and others
* with active or suspected malignant tumors, or with a previous history of malignant tumors, excluding skin basal cell carcinoma or cervical carcinoma in situ, within five (5) years before the screening
* with a history of major organ transplantation
* with a hypersensitive predisposition or a known history of serious allergy, especially to the investigational products and substances
* with a history of active alcohol or drug abuse within six (6) months before the screening
* pregnant women or lactating women rejecting or unable to discontinue nursing
* being unable to discontinue prohibited medications as defined by the protocol
* having previously participated in clinical studies of any other drugs within three (3) months before the screening
* being unable or unwilling to provide informed consent, or unable to follow the protocol requirements
* with any other conditions of ineligibility at the discretion of the investigators

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 371 (Actual)
Dates: Start 2017-06-07 (Actual); Primary Completion 2018-01-25 (Actual); Study Completion 2018-03-07 (Actual)

PRIMARY OUTCOMES:
Sustained virologic response at 12 weeks after end of treatment (SVR12) | 12 weeks after end of treatment
  Percentage of subjects with plasma HCV not detected or below the lower limit of quantitation (15 IU/mL)

SECONDARY OUTCOMES:
Sustained virologic response at 4 weeks after end of treatment (SVR4) | 4 weeks after end of treatment
  Percentage of subjects with plasma HCV not detected or below the lower limit of quantitation (15 IU/mL)
Rapid virologic response at 1 week after initiation of treatment (RVR1) | 1 week after initiation of treatment
  Percentage of subjects with plasma HCV not detected or below the lower limit of quantitation (15 IU/mL)
Rapid virologic response at 2 weeks after initiation of treatment (RVR2) | 2 weeks after initiation of treatment
  Percentage of subjects with plasma HCV not detected or below the lower limit of quantitation (15 IU/mL)
Rapid virologic response at 4 weeks after initiation of treatment (RVR4) | 4 weeks after initiation of treatment
  Percentage of subjects with plasma HCV not detected or below the lower limit of quantitation (15 IU/mL)
Rapid virologic response at 8 weeks after initiation of treatment (RVR8) | 8 weeks after initiation of treatment
  Percentage of subjects with plasma HCV not detected or below the lower limit of quantitation (15 IU/mL)
Rapid virologic response at 12 weeks after initiation of treatment (RVR12) | 12 weeks after initiation of treatment
  Percentage of subjects with plasma HCV not detected or below the lower limit of quantitation (15 IU/mL)

OTHER OUTCOMES:
Sustained virologic response at 24 weeks after end of treatment (SVR24) | 24 weeks after end of treatment
  Percentage of subjects with plasma HCV not detected or below the lower limit of quantitation (15 IU/mL)
Virologic breakthrough | 2, 4, 8 and 12 weeks after initiation of treatment
  Percentage of subjects with on-treatment re-detected plasma HCV RNA after HCV RNA below the lower limit of quantitation
Virologic relapse | 4,12 and 24 weeks after end of treatment
  Percentage of subjects with off-treatment re-detected plasma HCV RNA after end-of-treatment HCV RNA below the lower limit of quantitation

CONTACTS AND LOCATIONS:
Overall Officials: Junqi Niu, M.D., Principal Investigator — First Hospital of Jilin Univerisity; Lai Wei, M.D., Principal Investigator — Peking University People's Hospital
Locations (19):
- China (19):
  - Chinese PLA 302 Hospital, Beijing, Beijing Municipality
  - Capital Medical University Affiliated Beijing Youyi Hospital, Beijing, Beijing Municipality
  - Capital Medical University Affiliated Beijing You'an Hospital, Beijing, Beijing Municipality
  - Capital Medical University Affiliated Beijing Ditan Hospital, Beijing, Beijing Municipality
  - Chinese PLA Third Military Medical University First Affiliated Hospital, Chongqing, Chongqing Municipality
  - Chongqing Sanxia Central Hospital, Wanzhou, Chongqing Municipality
  - Sun Yat-sen University Affiliated Third University, Guangzhou, Guangdong
  - Guangzhou Municipal Eighth People's Hospital, Guanzhou, Guangdong
  - Liuzhou People's Hospital, Liuchow, Guangxi
  - He'nan Provincial Hospital of Infectious Disease (Zhengzhou Municipal Sixth People's Hospital), Zhengzhou, He'nan
  - Huazhong University of Science and Technology Affiliated Tongji Hospital, Wuhan, Hubei
  - Nanjing Municipal Second Hospital, Nanjing, Jiangsu
  - Jilin University First Hospital, Changchun, Jilin
  - Yanbian University Affiliated Hosptial, Yanbian, Jilin
  - Shenyang Municipal Sixth People's Hospital, Shenyang, Liaoning
  - Chinese PLA Fourth Military Medical University Tangdu Hospital, Xi'an, Shaanxi
  - Ji'nan Municipal Hospital of Infectious Disease, Ji'nan, Shandong
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Xinjiang Uygur Autonomous Region Traditional Chinese Medicine Hospital, Ürümqi, Xinjiang

IPD SHARING:
Plan to Share IPD: No
No IPD plan is included in the study protocol.